CLINICAL TRIAL: NCT02654275
Title: Effect of Proprioceptive Intervention Training on Power Capacity, Proprioceptive Ability and Technique of Young Swimmers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: Wingate College (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-15-HYMC
Record Dates: First submitted 2016-01-11; First posted 2016-01-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Injury Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Proprioceptive Intervention (Active Comparator): Strength training on a non-stable surface
  Interventions: Other: Proprioceptive Intervention
- No Proprioceptive Intervention (No Intervention): Conventional strength training

INTERVENTIONS:
Other: Proprioceptive Intervention
  Arms: Proprioceptive Intervention

SUMMARY:
Many children and adolescents who engage in swimming complain of shoulder pain during or after exercise. This pain may worsen and may lead to a decline in performance as well avoidance of swimming and lastly avoidance of any physical activity whatsoever. The aim of this study is to determine whether proprioceptive intervention training will effect the power capacity, proprioceptive ability and technique of young swimmers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Swim 3 times per week

Exclusion Criteria:

* Have not had orthopedic surgery
* No history of disease

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Change in proprioceptive ability | 8 weeks
  Biodex Device which measures joint proprioceptive ability, will measure the change before and after training

SECONDARY OUTCOMES:
Change in muscle strength | 8 weeks
  Biodex Device will measure the change in muscle isokinetic strength before and after training

CONTACTS AND LOCATIONS:
Overall Officials: Eias Kassem, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Wingate College, Netanya, Israel

IPD SHARING:
Plan to Share IPD: No